CLINICAL TRIAL: NCT03887104
Title: Data Collection of OCT and OCTA-based Ocular Measurements
Status: Completed | Type: Observational
Sponsor: Optovue (Industry)
Responsible Party: Sponsor
Other Study IDs: 200-53771
Record Dates: First submitted 2019-03-11; First posted 2019-03-22 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Eyes Without Ocular Pathology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

INTERVENTIONS:
Device: SD-OCT — Spectral Domain Optical Coherence Tomography for non-invasive, light-based, cross-sectional imaging of ocular structures

SUMMARY:
Data Collection of OCT and OCTA-based Ocular Measurements

DETAILED DESCRIPTION:
The purpose of this study is to collect measurements of anatomical structures of the posterior pole of the eye based on OCT scans in subjects without clinical signs of pathology.

ELIGIBILITY:
Inclusion Criteria:

* No glaucoma
* No retinal pathology
* No systemic disorders impacting the eye
* No ocular surgery or medical treatment of ocular condition

Exclusion Criteria:

* High IOP
* Poor vision
* Clinical findings consistent with pathology
* Unable to complete the study

Age Groups: Child, Adult, Older Adult
Study Population: Persons having eyes without ocular pathology
Sampling Method: Non-Probability Sample
Enrollment: 482 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2019-07-11 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Retinal thickness | Day 1
  micrometers

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Eye Care Center, Pomona, California
  - Eye Care Institute, Fort Lauderdale, Florida
  - IOVS, Newark, New Jersey
  - AMA Eye Physicians & Surgeons, Marysville, Ohio
  - College of Optometry, Tahlequah, Oklahoma